CLINICAL TRIAL: NCT04355260
Title: To Evaluate the Safety and Effectiveness Evaluation of Using Echocardiography-guided Liwen RF Radiofrequency Ablation System to Treat Hypertrophic Obstructive Cardiomyopathy
Brief Title: The Clinical Research of the Safety and Effectiveness Evaluation for Using Echocardiography-guided Liwen RF Radiofrequency Ablation System to Treat Hypertrophic Obstructive Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Hangzhou Nuo Cheng Medical Instrument Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Liu Liwen, MD.PHD., Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20192076-F-1
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-07

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Cardiomyopathy, hypertrophic;techniques; Treatment outcome
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertrophic Obstructive Cardiomyopathy (Experimental)
  Interventions: Procedure: Echocardiography-guided Radiofrequency ablation for Hypertrophic obstructive Cardiomyopathy (HOCM).

INTERVENTIONS:
Procedure: Echocardiography-guided Radiofrequency ablation for Hypertrophic obstructive Cardiomyopathy (HOCM). — Echocardiography-guided Radiofrequency ablation for Hypertrophic obstructive Cardiomyopathy (HOCM).

SUMMARY:
Objective to investigate the safety and effectiveness of Echocardiography-guided radiofrequency ablation in patients with Hypertrophic obstructive Cardiomyopathy (HOCM).

Percutaneous intramyocardial septal radiofrequency ablation (Liwen Procedure) is a safe and effective treatment approach for Hypertrophic obstructive Cardiomyopathy and results in sustained improvement in exercise capacity, persistent in reducing Left Ventricle Outflow Tract (LVOT) gradient, and sustained improvement in cardiac function.

In patients with disabling symptoms caused by Hypertrophic obstructive Cardiomyopathy (HOCM),Echocardiography-guided radiofrequency ablation could be a less invasive treatment option.

Percutaneous intramyocardial septal radiofrequency ablation (Liwen Procedure) is a new method for the diagnosis or treatment of heart disease by using a special diagnosis and treatment device to the heart target area under the guidance of image technology. The method breaks through the worldwide problem of the minimally invasive diagnosis and treatment of the myocardium on the beating heart, so as to avoid the X-ray radiation and contrast agent damage .

As a new pathway of cardiac disease intervention, Liwen Procedure can be used in congenital heart disease, myocardial biopsies, drug injection, cell implantation and instrument implantation in addition to Hypertrophic Cardiomyopathy and cardiac tumors. It has important clinical value and broad application prospect.

In this study, Liwen RF radiofrequency ablation system was used to treat HOCM , and evaluate its safety and effectiveness , in order to provide a new medical device for Liwen Procedure of HOCM.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has pressure gradient of left ventricular outflow tract (LVOT) ≥50 mmHg（with Systolic Anterior Motion）in the resting-state or after exercise stress test.
2. Subject with obvious clinical symptoms.
3. Subject with New York Heart Association (NYHA) cardiac function ≥ II grade.
4. Subject with adequate drug treatment is not effective or cannot tolerate side effects of the drug.
5. Subject was informed of the nature of the clinical study and agreed to participate in all the requirements of the clinical study, signed an informed consent form, and agreed to complete the following checks.

Exclusion Criteria:

1. Subject is pregnant, lactating, or planned to conceive during a clinical study.
2. Subject with Hypertrophic Non-obstructive Cardiomyopathy.
3. Subject with interventricular septal thickness ≥ 30mm.
4. Subject with Sudden Cardiac Death Index ≥ 10%.
5. Subject combined with other heart diseases requires surgical treatment.
6. Subject with heart failure(Defined as resting heart failure after intensive anti-heart failure therapy, left ventricular fraction of ejecting< 40%).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Main adverse event | 30 days
  Any instrument or surgery-related complications, including but not limited to death, emergency surgery, severe pericardial tamponade requiring pericardiocentesis or surgery, bleeding, surgery-related stroke.

SECONDARY OUTCOMES:
Instrument success | 30 days
  Radiofrequency ablation system instruments reach the desired treatment site and successfully complete ablation,and remove the system successfully.
Operation success | 90 days
  Improvement of LVOTG > 50% within 90 days after operation
No main adverse events related to instruments or surgery within 90 days of instrument use | 90 days
Life quality score of SF-36 | 90 days
  The life quality score of SF-36 was significantly improved after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Han C, Zhou M, Hu R, Wang B, Zuo L, Li J, Ta S, Hsi DH, Liu J, Wei L, Liu L. Trans-Septal Myocardial Biopsy in Hypertrophic Cardiomyopathy Using the Liwen Procedure: An Introduction of a Novel Technique. J Interv Cardiol. 2021 Feb 10;2021:1905184. doi: 10.1155/2021/1905184. eCollection 2021. PMID 33628143